CLINICAL TRIAL: NCT00641888
Title: Impact of Antiretroviral Therapy on Biomarkers of Inflammation Associated With Cardiovascular Risk
Brief Title: Impact of Antiretroviral Therapy on Cardiac Biomarkers
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: California HIV/AIDS Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: 200715922
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections
Keywords: Cardiovascular risk; Inflammatory biomarkers; Human immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 10 patients starting on non-nucleoside reverse transcriptase inhibitor based regimen. 5 women and 5 men.
- 2: 10 patients starting a protease inhibitor based regimen. 5 women and 5 men.

SUMMARY:
Cardiovascular risk appears to be linked to some degree with inflammation. HIV medications have been linked with cardiovascular risk. In this study we will be measuring levels of chemicals in the body associated with inflammation before and after starting HIV medications in patients with HIV. We hope to understand what happens to these chemicals once a patient with HIV is started on these medications to understand their role in cardiovascular risk.

DETAILED DESCRIPTION:
With the advent of antiretroviral therapy, death due to opportunistic diseases have seen a major decline among patients with HIV. However, several antiretroviral medications, in particular protease inhibitors (PI), have been associated with increased cardiovascular risk in large cohort studies. The role of inflammation in cardiovascular risk is currently being elucidated. High sensitivity C-reactive protein (hsCRP) has been identified as a strong independent predictor of cardiovascular disease among healthy individuals in several large cohort studies. Other inflammatory biomarkers such as serum amyloid A (SAA) and interleukin-6 (IL-6) have also been correlated with cardiovascular risk. Among patients with HIV, studies have revealed inappropriate immune activation with increased pro-inflammatory cytokines such as IL-6, IL-10, interferon-γ (IFN- γ), and tumor necrosis factor-α (TNF-α). The effects of this immune dysregulation and the impact of antiretroviral therapy on the cytokines and biomarkers associated with cardiovascular risk remain to be delineated.

Objective: Our aims are to characterize the levels of inflammatory biomarkers at the time of antiretroviral initiation, to define the time period over which the biomarkers change and stabilize, and to determine if the type of antiretroviral drug class used has an impact on the rate of alteration of these biomarkers. Given the disparate cardiovascular risk between women and men of similar age groups, we will study the additional impact of gender on these biomarkers. We will also explore whether there is a correlation between change of CD4 T-lymphocyte counts and the response of the biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a CD4 count between 200-400 planning on initiating antiretrovirals.

Exclusion Criteria:

* Pregnancy,
* Recent discontinuation of an antiretroviral within the past 30 days,
* Active intravenous drug use,
* Acute febrile illness with temperature > 100 F,
* Diagnosis or symptoms of acute infection within the past 30 days,
* Opportunistic infection or surgical procedure within the past 60 days,
* Myocardial infarction within the last 30 days,
* Renal disease (CKD Stages 3-5), and
* Unstable liver disease.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an HIV clinic and an infectious diseases clinic affiliated with a tertiary care hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Archana Maniar, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States